CLINICAL TRIAL: NCT06870214
Title: ''Investigation of the Effect of Benson Relaxation Technique Applied to Pregnant Women on Fear of Childbirth, Anxiety and Stress Levels of Pregnant Women''
Brief Title: Benson Relaxation Technique and Stress in Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Sümeyye BAL, Lecturer Ph. D., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-930
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Stress; Relation, Interpersonal
MeSH Terms: conditions — Anxiety Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relaxation group (Experimental): They will be interviewed according to the inclusion criteria and exclusion criteria, and they will be informed about the study and their consent will be obtained, the participant information form and depression form will be filled, a pre-test will be performed and the communication will be completed. Their numbers will be taken.
  The intervention group will be given a 1-hour Benson relaxation technique every week for 4 weeks. Participants will be asked to do relaxation exercises for 10 to 15 minutes twice a day, in the morning and evening, for 1 month. A phone number will be provided for patients to call if they have questions. In addition, the researcher will call the women in the intervention group every week to follow up on the relaxation process and answer questions.
  The researcher will contact the experimental group by phone. He/she will introduce himself/herself and final tests will be conducted after 4 weeks.
  Interventions: Other: relaxation
- control group (No Intervention): **"Routine nursing care will be provided."**

INTERVENTIONS:
Other: relaxation — Women in the 3rd trimester will receive routine care only.
  Other Names: control group
  Arms: relaxation group

SUMMARY:
The aim of this study is to determine the effect of the Benson Relaxation Technique applied to pregnant women on their fear of birth, anxiety and stress levels.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of the Benson Relaxation Technique applied to pregnant women on their fear of birth, anxiety and stress levels.

Hypotheses ; H0-1: Benson relaxation technique applied to pregnant women has an effect on childbirth.

H1-1: Benson relaxation technique applied to pregnant women has no effect on childbirth.

H0-2: Benson relaxation technique applied to pregnant women has no effect on anxiety.

H1-2: Benson relaxation technique applied to pregnant women has an effect on anxiety.

H0-3: Benson relaxation technique applied to pregnant women and their partners has no effect on stress.

H1-3: Benson relaxation technique applied to pregnant women and their partners has an effect on stress The study will be conducted on two different groups. The application will be a 1-hour Benson relaxation technique applied to pregnant women in the third trimester every week for 4 weeks. Participants will be asked to do relaxation exercises twice a day, morning and evening, for 10 to 15 minutes for 1 month. A phone number that patients can call with questions will also be provided. In addition, the researcher will call the women in the intervention group every week to follow up on the relaxation process and answer questions.

After the women are evaluated in terms of eligibility criteria for the study, information about the study will be provided to the women who are eligible and written informed consent will be obtained from the women who accept. The random distribution of the women to the study groups will be carried out using the Block Randomization method. The following applications will be applied to the groups.

The researcher will contact the experimental group by phone. The application will end after 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those who are in their 28th-38th weeks of pregnancy,
* People with mental illness,
* People who have Anxiety disorder,
* People with hearing loss;
* People who have no experience of using relaxation methods in the past,
* People who have not used herbal or medical sedatives

Exclusion Criteria:

* Those who do not want to participate in the intervention,
* Those who have a termination of pregnancy during the intervention,
* Those who have a risky pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
1.Change in anxiety | immediately intervention 4 weeks later
  Beck Anxiety Inventory scale (BAI). The BAI measures only the frequency of anxiety symptoms in detail. It is a Likert-type self-assessment scale comprised of 21 items scored between 0 and 3. The higher the total score, the higher the anxiety experienced by the person (minimal: 0-7, mild: 8-15, moderate:16-25, and severe: 26-63 points). 18 The Turkish validity and reliability of the BSI has been reported by Ulusoy et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No